CLINICAL TRIAL: NCT00394550
Title: Treatment of Children With Obstructive Sleep Apnea and Laryngomalacia: the Role of Laser Supraglottoplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient institutional support
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Bruce Matt, Associate Professor, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1011003593
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Sleep Apnea, Obstructive; Respiration Disorders
Keywords: laryngomalacia; supraglottoplasty; Tonsillectomy; Adenoidectomy; obstructive sleep apnea; Laser; Polysomnogram; airway obstruction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Respiration Disorders; Laryngomalacia; Airway Obstruction | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): If laryngomalacia is found, then in the control group, no supraglottoplasty will be performed. Only the tonsils and adenoids will be removed.
- Treatment (Experimental): If laryngomalacia is found, then in the Treatment group, a supraglottoplasty with laser will be performed, as well as removal of the tonsils and adenoids.
  Intervention: supraglottoplasty with laser
  Interventions: Procedure: supraglottoplasty with laser

INTERVENTIONS:
Procedure: supraglottoplasty with laser — Polysomnogram, fiberoptic flexible laryngoscopy, adenotonsillectomy, direct laryngoscopy, bronchoscopy, laser supraglottoplasty, general anesthesia, a proton-pump inhibitor ibuprofen, acetaminophen with codeine without alcohol, or other narcotic containing medication, antibiotic, possible use of other analgesics per anesthesia None of these procedures are "new" or experimental. Our investigation pertains to a broader use of the laser supraglottoplasty to include children with obstructive sleep apnea and laryngomalacia, as opposed to the more traditional use of laser supraglottoplasty for only severe laryngomalacia in young children
  Arms: Treatment
Procedure: supraglottoplasty with laser — laser excision of laryngomalacia (floppy tissue) on one side of the supraglottis
  Arms: Treatment

SUMMARY:
This is a research study of the effect of treating laryngomalacia (floppiness of tissue on top of the voice box that can possibly block breathing) found in association with obstructive sleep apnea (blockage of breathing while sleeping).

The purpose of this study is to determine which is the best treatment for children with obstructive sleep apnea and laryngomalacia: adenotonsillectomy alone or adenotonsillectomy with laser supraglottoplasty (removal of tissue on top of the voice box to open the airway).

DETAILED DESCRIPTION:
If you agree to have your child be in the study, you will do the following things:

you are consenting to your child having the adenoid (tissue similar to lymph nodes, found in the back of the throat) and tonsils removed (if not previously performed), direct laryngoscopy (looking in the throat) and bronchoscopy (inspection of the lungs with a long tube-like device down the throat), and randomization (½ will be treated further, ½ will be observed) into treatment and no-treatment arms if your child is diagnosed with laryngomalacia. After starting general anesthesia (putting patient to sleep for procedure), the surgeon will perform direct laryngoscopy (look at the throat and voice box) and bronchoscopy (look at the entrance to the lungs [trachea or windpipe]). If your child is diagnosed with laryngomalacia (flopping of the tissue around the voice box, potentially causing obstruction or blockage), 50% will undergo a further treatment (laser supraglottoplasty, or removal of tissue at the entrance of the voice box) and 50% will be observed. The decision to treat or not treat will be random, as is customary for prospective research trials. All children (both treatment arms will receive a 3 week treatment of a medicine (a proton pump inhibitor) to reduce the level of stomach acid and prevent potential exposure of the larynx (voice-box) to stomach acid. If your child does not have laryngomalacia, no further treatment on the larynx (voice-box) will be performed. Next, adenotonsillectomy will be performed as is common for the Otolaryngologist performing the procedure. Postoperatively, a sleep study will be performed (identical to the preoperative study) ideally 3-6 months after surgery, (but up to one year after) to monitor your child's progress. Additional laboratory tests or drawing of blood is not routine in this procedure, but may be performed as dictated by your child's medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* 1 year old to 18 years of age, clinical signs or symptoms of obstructive sleep apnea (snoring, witnessed apneas, daytime somnolence, restless sleeping, or cyanosis), abnormal polysomnogram (mild, moderate, or severe OSA) including CO2 measures, failed or refused trial of CPAP, or not recommended by their pulmonologist or primary care doctor.

Exclusion Criteria:

* prior laser supraglottoplasty, prior adenoidectomy prior tonsillectomy, stridor with cyanosis or apnea, severe respiratory distress, recurrent pneumonia (x3), Laryngeal cyst, vocal cord (VC) Paralysis, airway vascular malformation, neoplasm, subglottic hemangioma, paradoxical vocal cord (VC) motion, posterior glottic stenosis, glottic webs, discoordinate pharyngolaryngomalacia, or refusal to participate.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
as measured by overnight polysomnogram: | within one year of operation
Changes in minimum oxygen saturation | within one year of operation
Changes in Respiratory Disturbance index | within one year of operation
Changes in peak end-tidal carbon dioxide(CO2) level | within one year of operation
Changes in mean end-tidal carbon dioxide(CO2) level | within one year of operation

SECONDARY OUTCOMES:
overall category of airway obstruction on polysomnogram (e.g. normal, mild, moderate, severe obstructive sleep apnea) | within one year of operation

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H. Matt, MD, MSc, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Childrens' Hospital, Indianapolis, Indiana, United States